CLINICAL TRIAL: NCT03771950
Title: Early Team Based Neuro-rehabilitation After Traumatic Brain Injury - a Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Alingsas hospital emergincy section (Unknown); Narhalsan primary care rehabilitation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 470-18
Record Dates: First submitted 2018-11-27; First posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Traumatic Brain Injury; Concussion, Brain
Keywords: rehabilitation
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: After screening for eligibility, fulfilling inclusion criteria and consenting to participation the baseline assessment will be conducted by an OT at enrolment. After this the patients will be randomised either to the intervention or control group in using lots in sealed envelopes based on a computer generated group allocation. The lots are kept in sealed envelopes prepared by a person not involved in the study. An OT will open the envelope and inform the patient about group allocation. All care providers will be blinded for baseline and post-test outcomes. A research co-worker who are involved in data management will be blinded for group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Early team based neuro-rehabilitation after Traumatic Brain Injury
  Interventions: Behavioral: Early team based neuro-rehabilitation
- Control group (No Intervention): Treatment as usual.

INTERVENTIONS:
Behavioral: Early team based neuro-rehabilitation — A structured interview will be made by OT about activity level, and an examination of the patients bodily and neurological symptoms will be made by PT. Based on this result a rehabilitation plan is established consisting of the patient's goals, and the purpose that the patient shall be as active as possible without triggering symptoms. An individual exercise program is prescribed. Between each appointment the patient will have personal tasks to accomplish with the purpose of being active based on symptoms and the adaptation to the current level of energy. The perceived symptoms will be logged. A week-schedule will be created in the purpose of helping the patient to a balanced activity level in relation to their current capacity. The PT assesses physical activity level and reactions to physical strain. Adaptations are made to the exercise program and advice is given on physical activity and exercises. When appropriate OT advices about returning to work and adaptations concerning work.
  Arms: Intervention group

SUMMARY:
The aim is to evaluate the study design, procedure and measurements in a randomised controlled pilot study.

DETAILED DESCRIPTION:
Despite that mild traumatic brain injury (mTBI) is a common condition managed in various healthcare settings, early team based neurorehabilitation (TbNR) in post-concussion syndrom (PCS) is sparely investigated. Therefore we aim to design a high quality randomised controlled study (RCT) investigating the effect of early TbNR in PCS. Prior this RCT a pilot study will be conducted with the aim to evaluate the study design, procedure and measurements.

Method:

Thirty consecutive patients visiting Alingsås hospital emergency department due to head injury caused by fall, trauma to the head, traffic accident or abuse, and diagnosed with brain concussion (ICD10 S060, S0600) for the first time or after repeated trauma, will be asked to participate in the study. The patient will receive a written study information when discharged, and asked if an occupational therapist can contact the patient by phone for further information and screening questions 14 days after trauma. If the patient meet the inclusion criteria and wish to participate in the study a written informed consent will be obtained.

Test procedure:

A structured interview and the assessment described below will be performed at baseline 3-4 weeks after the trauma and after 16 weeks by an occupational therapist. Participant's characteristics such as age, gender, work ability, education, social status, previous trauma to the head and known comorbidity are collected. The classification of the mTBI will be collected from the patients' medical journal, as well as the result and time of the CT examination if it has been performed. Information about previous sick leave will be collected from the Swedish health insurance office. The number of visits to the occupational therapist (OT) and the physiotherapist (PT) will be recorded from the participant's medical journal.

Study protocol In this pilot study we plan to evaluate broadly as the persons with mTBI may suffer from a complex symptomatology, and the causes of persisting symptoms are unclear.

The following data will be collected:

* The number of patients who meet the inclusion criteria.
* The number of patients consenting participation in the study.
* The number of patients completing questionnaires at baseline and post-test.
* The number of patients who participate in the intervention.

Randomisation:

After screening for eligibility, fulfilling inclusion criteria and consenting to participation the baseline assessment will be conducted by an OT at enrolment. After this the patients will be randomised either to the intervention or control group in using lots in sealed envelopes based on a computer generated group allocation. The lots are kept in sealed envelopes prepared by a person not involved in the study. An OT will open the envelope and inform the patient about group allocation. All care providers will be blinded for baseline and post-test outcomes. A research co-worker who are involved in data management will be blinded for group allocation.

Interventions:

The patients randomised to the intervention group (n=15) will be treated by the PT and OT in TbNR. At the first visits a medical history will be taken, there after a structured interview will be made by the OT about activity level, and an examination of the patients bodily and neurological symptoms will be made by the PT. Based on this result a TbNR a rehabilitation plan is established consisting of the patient's goals, and the purpose that the patient shall be as active as possible without triggering symptoms. An individual exercise program is prescribed. Number of visits to TbNR will depend on the individual need for rehabilitation.

Between each appointment with TbNR, the patient will have personal tasks to accomplish with the purpose of being active based on symptoms and the adaptation to the current level of energy. Information about underlying causes of perceived symptoms will be present at the visits, and the patient will be given help to analyze the tasks that has been performed during the past week. The perceived symptoms will be logged in an activity log including estimation of fatigue and headache. A week-schedule will be created in the purpose of helping the patient to a balanced activity level in relation to their current capacity.

The PT assesses physical activity level and reactions to physical strain. Adaptations are made to the exercise program and advice is given on physical activity and exercises. When appropriate the OT advices about returning to work and adaptations concerning work.

Control:

Participants will be treated as usual, which is that they can search health care by themself.

Statistics:

Ratio and interval data are presented as mean ± 1 standard deviation (SD), ordinal data are presented as median, and 25th and 75th percentile, nominal data are presented in absolute and relative numbers.

Change between baseline and post-test will be analyzed for each outcome measure and between the groups. Depending if the data are normal distributed or not parametric or non-parametric tests will be used for differences between group.

Effect sizes and 95% confidence intervals will be calculated. Cohen's d will be used to estimate the effect size using mean difference between groups and pooled standard deviation of the mean differences. The magnitude of effect size will be considered small for d = 0.2 - 0.49, medium for d = 0.5-0.79, and large for d = 0.8-1.1 (16).

Odds ratio will be used to estimate effect size for binary dependent variable using logistic regression. Linear regression analysis will be used for change of outcome measurements adjusting for gender, number of head trauma and if the injury has been caused by another person or not. The Statistical Package for Social Science (SPSS) for Windows, Version 22.0, 2013. IBM Corp, Armonk, NY: USA will be used for statistical analyses. A p-value < 0.05 is considered statistical significant.

Sample size:

In the planned pilot study 30 participants will be enrolled. This sample size is considered to be sufficient to analyze effect size for the included outcome measurements which will be used for planning the full-scale randomized controlled study involving more emergency hospitals and neuro teams.

ELIGIBILITY:
Inclusion criteria:

* Head injury for the first time or repeated trauma.
* Diagnosed with brain concussion (ICD10 S060, S0600) by a physician.
* Persistent symptoms after mTBI or decreased activity level at time for inclusion.

Exclusions criteria:

* No remaining symptoms after mTBI at time for inclusion.
* Returned to previous activity daily living level as before trauma.
* Other serious illness.
* Unwillingness to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Numbers of patients who meet the inclusion criteria and accept participation in the study? | 16 weeks after trauma
  Count how many of the patients want to participate in the study

SECONDARY OUTCOMES:
Numbers of participants who respond to the included measurements? | 16 weeks after trauma
  Count the number
Numbers of participants who complete post-test? | 16 weeks after trauma
  Count the number
Rivermead post-concussion symtoms questionnaire (Swedish version) (RPQ) | Effect size of change from baseline to 16 weeks after trauma
  A valid, reliable and established measurement of self-perceived symptoms after brain concussion. The measurement consists of 16 items concerning perceived headache, vertigo, nausea, sensitivity to sound, sleeping disorders, fatigue, irritability, depression, frustration, poor memory, poor concentration, longer time to think, blurred vision, sensitivity to light, double vision and restlessness the past 24 hours compared to before the head injury. The symptoms are assessed on a 5-pointscale: never had symptom (category 0), had symptoms but they resolved (category 1), had moderate problems with symptom (category 2), having moderate problems with symptom (category 3), having severe problem with symptom (category 4)
Multidimensional Fatigue Inventory (MFI) | Effect size of change from baseline to 16 weeks after trauma
  A valid and reliable measurement consisting of 20 items to measure fatigue. Various dimensions are estimated such as general fatigue, physical fatigue, decreased activity, reduced motivation and mental fatigue.
Activity level is measured with GAP in everyday activity. | Effect size of change from baseline to 16 weeks after trauma
  GAP measures participation by capturing the difference between what the patient wants to perform and actually performs. The measure consists of 30 items and the participant answers yes or no if the person performs the activity, and yes or no if the person wants to perform it.
Leisure Time Physical Activity Instrument (LTPI) (Swedish version) | Effect size of change from baseline to 16 weeks after trauma
  Captures the participant physical activity level: sedentary, light activity (does not increase respiratory rate), moderate activity (increased respiratory rate and increased body temperature), high activity level (significantly increases respiratory rate and body temperature)
Sleep quantity is measured by two questions: | Effect size of change from baseline to 16 weeks after trauma
  "Do you think that you get enough sleep?". Sleep quality is measured by the question: "Considering all, how do you think that you sleep?" The participants answers the questions on a four-grade-scale: the higher number-the better
RAND-36 | Effect size of change from baseline to 16 weeks after trauma
  Consists of 36 items that measure health-related quality of life comprising eight subscales ranging from 0-100. The subscales are physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional and mental health
Hospital Anxiety and Depression Scale (HADS Swedish version) | Effect size of change from baseline to 16 weeks after trauma
  A self-evaluation measure of anxiety and depression in patients in somatic health care. HADS consists of 14 statements (0-21) for each part: HADS-anxiety and HADS-depression. Higher score indicate more server anxiety and depression.
Gender, male and female | Relation between gender and change from baseline to 16 weeks after trauma in the outcomes measurements RPQ, MFI, LTPAI,GAP, Sleep, HADS.
  Gender will be collected from the participant medical record at baseline
Number of head trauma | Relation between number of head trauma and change from baseline to 16 weeks after trauma in the outcomes measurements RPQ, MFI, LTPAI,GAP, Sleep, HADS.
  Number of head trauma will be collected from the participants medical record at baseline
Trauma caused by another person or not (yes/no) | Relation between trauma caused by another person or not and change from baseline to 16 weeks after trauma in the outcomes measurements RPQ, MFI, LTPAI,GAP, Sleep, HADS.
  Information about if trauma is caused by another person or not, will be collected from the participants medical record at baseline
Self-reported comorbidity | Relation between self-reported comorbidity and change from baseline to 16 weeks after trauma in the outcomes measurements RPQ, MFI, LTPAI,GAP, Sleep, HADS.
  Information about comorbidity will be collected in a structured interview at baseline
Computer Tomografi (CT) assessment | Relation between CT assessment and change from baseline to 16 weeks after trauma in the outcomes measurements RPQ, MFI, LTPAI,GAP, Sleep, HADS.
  If Computer Tomografi (CT) assessment was used be collected from the participants medical record at baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Narhalsan Sorhaga Rehabmottagning, Alingsås, Vasta Gotaland, Sweden

REFERENCES:
- [Background] Lannsjo M, af Geijerstam JL, Johansson U, Bring J, Borg J. Prevalence and structure of symptoms at 3 months after mild traumatic brain injury in a national cohort. Brain Inj. 2009 Mar;23(3):213-9. doi: 10.1080/02699050902748356. PMID 19205957
- [Background] Lundin A, de Boussard C, Edman G, Borg J. Symptoms and disability until 3 months after mild TBI. Brain Inj. 2006 Jul;20(8):799-806. doi: 10.1080/02699050600744327. PMID 17060147
- [Background] Belmont A, Agar N, Azouvi P. Subjective fatigue, mental effort, and attention deficits after severe traumatic brain injury. Neurorehabil Neural Repair. 2009 Nov;23(9):939-44. doi: 10.1177/1545968309340327. Epub 2009 Jul 2. PMID 19574545
- [Background] Ponsford J, Cameron P, Fitzgerald M, Grant M, Mikocka-Walus A. Long-term outcomes after uncomplicated mild traumatic brain injury: a comparison with trauma controls. J Neurotrauma. 2011 Jun;28(6):937-46. doi: 10.1089/neu.2010.1516. Epub 2011 May 25. PMID 21410321
- [Background] Middleboe T, Andersen HS, Birket-Smith M, Friis ML. Minor head injury: impact on general health after 1 year. A prospective follow-up study. Acta Neurol Scand. 1992 Jan;85(1):5-9. PMID 1546534
- [Background] Ziino C, Ponsford J. Selective attention deficits and subjective fatigue following traumatic brain injury. Neuropsychology. 2006 May;20(3):383-90. doi: 10.1037/0894-4105.20.3.383. PMID 16719631
- [Background] Cassidy JD, Cancelliere C, Carroll LJ, Cote P, Hincapie CA, Holm LW, Hartvigsen J, Donovan J, Nygren-de Boussard C, Kristman VL, Borg J. Systematic review of self-reported prognosis in adults after mild traumatic brain injury: results of the International Collaboration on Mild Traumatic Brain Injury Prognosis. Arch Phys Med Rehabil. 2014 Mar;95(3 Suppl):S132-51. doi: 10.1016/j.apmr.2013.08.299. PMID 24581902
- [Background] Lannsjo M, Borg J, Bjorklund G, Af Geijerstam JL, Lundgren-Nilsson A. Internal construct validity of the Rivermead Post-Concussion Symptoms Questionnaire. J Rehabil Med. 2011 Nov;43(11):997-1002. doi: 10.2340/16501977-0875. PMID 22031345
- [Background] Smets EM, Garssen B, Bonke B, De Haes JC. The Multidimensional Fatigue Inventory (MFI) psychometric qualities of an instrument to assess fatigue. J Psychosom Res. 1995 Apr;39(3):315-25. doi: 10.1016/0022-3999(94)00125-o. PMID 7636775
- [Background] Mannerkorpi K, Hernelid C. Leisure Time Physical Activity Instrument and Physical Activity at Home and Work Instrument. Development, face validity, construct validity and test-retest reliability for subjects with fibromyalgia. Disabil Rehabil. 2005 Jun 17;27(12):695-701. doi: 10.1080/09638280400009063. PMID 16012062
- [Background] Akerstedt T, Knutsson A, Westerholm P, Theorell T, Alfredsson L, Kecklund G. Sleep disturbances, work stress and work hours: a cross-sectional study. J Psychosom Res. 2002 Sep;53(3):741-8. doi: 10.1016/s0022-3999(02)00333-1. PMID 12217447
- [Background] Hays RD, Morales LS. The RAND-36 measure of health-related quality of life. Ann Med. 2001 Jul;33(5):350-7. doi: 10.3109/07853890109002089. PMID 11491194
- [Background] Lisspers J, Nygren A, Soderman E. Hospital Anxiety and Depression Scale (HAD): some psychometric data for a Swedish sample. Acta Psychiatr Scand. 1997 Oct;96(4):281-6. doi: 10.1111/j.1600-0447.1997.tb10164.x. PMID 9350957
- [Background] Sawilowsky S. New Effect Size Rules of Thumb. Journal of Modern Applied Statistical Methods [Internet]. 2009 Nov 1;8(2). Available from: http://digitalcommons.wayne.edu/jmasm/vol8/iss2/26 OCH Cohen J. Statistical power analysis for the behavioral sciences. Second edition. Hillsdale: Routlegde; 1988.